CLINICAL TRIAL: NCT07197528
Title: Effectiveness of Precision Rehabilitative Exercise Training on Sarcopenia, Joint Range of Motion, Cognitive Function, Activities of Daily Living, Quality of Life, and Mood Status in Elderly Residents of Long-Term Care Facilities
Brief Title: Effectiveness of Smart-Assisted Rehabilitation Exercise Training on the Physical and Mental Health of Older Adults in Long-Term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, ZENG SIOU RONG, Co-Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A202405161
Record Dates: First submitted 2025-07-23; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia in Elderly; Rehabilitation Exercise; Long Term Care
Keywords: sarcopenia; elderly; rehabilitation; Long Term Care
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Experimental: Intervention Group Participants will receive a 12-week exercise training program using the smart-assisted rehabilitation system "KNEESUP." The training includes progressive resistance exercises tailored to individual functional abilities, conducted three times per week with two sessions per day. The system provides real-time monitoring, feedback, and remote adjustments by rehabilitation specialists.
  Interventions: Behavioral: Experimental Arm：Smart-assisted rehabilitation exercise system Control Arm：Usual care or routine physical activity
- Control Group (No Intervention): Participants will receive usual care, including standard daily activities and routine rehabilitation therapies provided by the long-term care facility, without use of the smart-assisted rehabilitation system.

INTERVENTIONS:
Behavioral: Experimental Arm：Smart-assisted rehabilitation exercise system Control Arm：Usual care or routine physical activity — Interventions
  Behavioral: Smart-assisted rehabilitation exercise system ("KNEESUP") A wearable smart-assisted rehabilitation system providing personalized, progressive lower limb resistance training for elderly residents with sarcopenia in long-term care institutions. The system includes real-time monitoring, feedback, and remote adjustment by rehabilitation specialists. Unlike traditional programs, it integrates sensor technology to track knee joint angles and exercise performance, enabling precise and adaptive training.
  Other: Usual care / routine physical activity Participants follow standard daily activities and rehabilitation provided by the long-term care facility, without the smart-assisted rehabilitation system.
  Arms: Intervention Group

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness of a smart-assisted rehabilitation system on the physical and mental health of elderly residents in long-term care facilities through exercise training.

The specific aim of this study is to investigate the effects of a 12-week exercise training program using a smart-assisted rehabilitation system on sarcopenia, joint range of motion, cognitive function, activities of daily living, functional status, quality of life, and emotional well-being among institutionalized older adults.

Participants will be divided into an experimental group and a control group for comparison to assess whether the intervention improves outcomes such as sarcopenia, joint mobility, cognitive function, daily living abilities, overall functional status, quality of life, and emotional state.

Participants in the experimental group will receive the "KNEESUP" smart medical rehabilitation system, provided by a co-investigator. A rehabilitation physician will design an individualized, progressive exercise program. The intervention is planned for 12 weeks, with a frequency of 3 days per week, 2 sessions per day, totaling 72 sessions.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effectiveness of a 12-week exercise intervention using an intelligent rehabilitation assistance system (KNEESUP) in improving the physical and mental health of institutionalized older adults with sarcopenia in long-term care facilities.

With the rapid aging of the population, long-term care institutions have become crucial in supporting the quality of life for older adults. Residents in these settings often face compounded challenges, including chronic illnesses, reduced physical function, cognitive decline, and psychosocial issues such as loneliness and depression. These conditions increase the burden on healthcare systems and care staff. While exercise interventions are known to be effective in promoting physical and mental well-being in older adults, traditional standardized programs may lack individualization and precision.

This study introduces a smart rehabilitation system that combines wearable technology and personalized exercise prescriptions designed by a physical medicine and rehabilitation physician. The system allows real-time monitoring and feedback, which enhances safety, motivation, and adherence. The intervention aligns with trends in post-pandemic digital health solutions and aims to integrate medical technology into routine elder care.

Study Design A randomized controlled trial will be conducted. Eligible participants (aged ≥65 with sarcopenia, able to stand with assistance or walk with/without aid, and cognitively intact) will be randomly assigned to either an intervention or control group in a 1:1 ratio. The sample size was calculated using G*Power, estimating 42 participants to account for a 20% dropout rate.

Intervention group: Receives a 12-week progressive resistance training program using the KNEESUP smart rehabilitation system. Training will occur 3 times per week, twice per day, totaling 72 sessions. Exercises include lower-limb strengthening through progressive stages (bed, seated, and standing), designed by a team of multidisciplinary experts and monitored via wearable sensors.

Control group: Continues routine care and usual physical activity without additional intervention.

Outcome Measures

Participants will be assessed pre- and post-intervention on the following variables:

Sarcopenia indicators: Grip strength, limb circumference

Joint range of motion: Measured with goniometer (upper limbs) and the KNEESUP system (lower limbs)

Cognitive function: Short Portable Mental Status Questionnaire (SPMSQ)

Daily living function: Barthel Index

Functional status: Comprehensive Geriatric Assessment (CGA)

Quality of life: WHOQOL-BREF (Taiwan version)

Emotional state: Geriatric Depression Scale (GDS-15)

Basic demographic and lifestyle data: Age, sex, education, comorbidities, social support, and physical activity habits

Statistical Analysis Data will be analyzed using SPSS. Descriptive statistics (mean, SD, percentage) and inferential statistics (independent t-tests, chi-square tests, ANOVA, and generalized estimating equations [GEE]) will be used to assess within-group and between-group differences, and group × time interaction effects. Significance is set at α = 0.05.

Data Management and Confidentiality All data will be anonymized. Paper and electronic data will be securely stored and encrypted. Data will be destroyed 5 years after study completion. Only authorized personnel will have access.

Ethical Considerations The study has IRB approval and informed consent will be obtained from all participants or their legal guardians. Risks (e.g., muscle soreness or fatigue) will be mitigated with one-on-one supervision. Emergency procedures and referral systems are in place if adverse events occur.

Expected Impact This study is expected to provide evidence supporting the feasibility and effectiveness of smart rehabilitation systems in long-term care. It may serve as a model for future eldercare strategies, inform policy, and contribute to the development of precision geriatric rehabilitation approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 65 years or older residing in long-term care facilities and diagnosed with sarcopenia, defined as:

   * Handgrip strength: <28 kg for males or <18 kg for females, or
   * Calf circumference (10 cm below the knee): <34 cm for males or <33 cm for females.
2. Able to stand with assistive devices (e.g., walker), transfer from bed to chair using a wheelchair, or ambulate independently.
3. Clear consciousness, able to communicate, and able to provide informed consent.
4. Willing to participate and comply with the exercise intervention.

Exclusion Criteria:

1. Impaired consciousness.
2. Unsuitable for wearing the device due to any leg-related medical condition.
3. Unable to perform aerobic or resistance training due to neurological or musculoskeletal disorders.
4. History of head injury resulting in cognitive impairments such as memory or attention deficits.
5. Assessed by a rehabilitation specialist as having absolute or relative contraindications to exercise training, such as:

   * Severe myocardial ischemia
   * Myocardial infarction within the past 6 months
   * Unstable angina
   * Uncontrolled arrhythmias causing symptoms or hemodynamic instability
   * Severe aortic valve stenosis
6. Deemed unsuitable to participate in the study by a rehabilitation specialist due to conditions such as end-stage renal disease requiring dialysis, terminal cancer, or ongoing chemotherapy/radiation therapy.
7. Diagnosed with depression or experienced major life events in the past six months.
8. Fracture, sports injury of the limbs, stroke, dementia, or other major illness within the past six months.
9. Individuals with infectious disease risks.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-05-18 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
Upper limb grip strength | From enrollment to the end of treatment at 12 weeks
  Grip strength was assessed using the Jamar 5030J1 analog dynamometer. Participants performed two consecutive grip tests with their dominant hand, and the highest value from the two trials was recorded. Grip strength values indicating possible sarcopenia are <28 kg for males and <18 kg for females.
Calf and arm circumferences | From enrollment to the end of treatment at 12 weeks
  Calf and arm circumferences will be measured using a tape measure.
  Calf circumference: measured in a seated position at the widest part of the calf. A value <34 cm for males and <33 cm for females indicates risk of sarcopenia.
  Arm circumference: measured at the midpoint of the non-dominant upper arm. A value ≤28.6 cm for males and ≤27.5 cm for females indicates risk of sarcopenia.

SECONDARY OUTCOMES:
Range of Motion | From enrollment to the end of treatment at 12 weeks
  For the upper limbs, joint angles of the shoulder and elbow were measured using a traditional goniometer. For the lower limbs, the hip and knee joints were measured using the "KNEESUP" device and its associated application. After turning on the "KNEESUP" device, it connects to a smartphone via Bluetooth, allowing the sensor to detect the participant's lower limb movements, knee flexion angles, the time taken to complete movements, and the accuracy of the movements. These data are transmitted to the app for analysis.
Cognitive Function | From enrollment to the end of treatment at 12 weeks.
  This study uses the Short Portable Mental Status Questionnaire (SPMSQ) to assess the cognitive function of elderly participants. The questionnaire covers six dimensions: consciousness, memory, orientation, attention, thinking, and general knowledge, with a total of 10 items.
Activities of Daily Living (ADL) | From enrollment to the end of treatment at 12 weeks.
  This study uses the Barthel Index to assess the basic self-care abilities of elderly individuals in the community and all care facilities. The main assessment items include seven self-care abilities and three mobility skills, totaling 10 evaluation items. The scores are categorized as follows: complete dependence (0-20 points), severe dependence (21-60 points), moderate dependence (61-90 points), mild dependence (91-99 points), and complete independence (100 points).
Quality of Life Assessed Using WHOQOL-BREF | From enrollment to the end of treatment at 12 weeks.
  The Taiwan version of the WHOQOL-BREF consists of 28 items, including two global items assessing overall quality of life and general health, and 26 items across four domains: physical health, psychological health, social relationships, and environment. Each item uses a 5-point Likert scale. Negatively phrased items are reverse-coded. Higher scores reflect better perceived quality of life. This version includes two additional culturally relevant items developed for the Taiwanese population. Domain reliability ranges from Cronbach's α = 0.70 to 0.77.
Depressive Symptoms Assessed Using the Chinese Version of the Geriatric Depression Scale-15 (CT-GDS-15) | From enrollment to the end of treatment at 12 weeks.
  Emotional status will be assessed using the Chinese-Translated Geriatric Depression Scale-15 (CT-GDS-15), a 15-item screening tool for depressive symptoms in older adults. Items are answered with "yes" or "no" and scored 0-15. Higher scores indicate more severe depressive symptoms. A score of 0-6 suggests normal emotional status, 7-10 indicates mild to moderate depression, and ≥11 suggests severe depression requiring further evaluation. The scale has a reported sensitivity of 72% and specificity of 57% based on DSM-III criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Banqiao Veterans Home of Veterans Affairs Council, R.O.C., New Taipei City, Banqiao Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No